CLINICAL TRIAL: NCT05758051
Title: Management of Slipped Capital Femoral Epiphysis (SCFE) on Top of Fixed Fracture Neck of Femur Case Report.
Acronym: SCFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hesham Mohamed Elbaseet, Principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCFENOF
Record Dates: First submitted 2023-02-05; First posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Slipped Capital Femoral Epiphysis
Keywords: Slipped capital femoral epiphysis; SCFE; coxa vara; fracture neck of femur
MeSH Terms: conditions — Slipped Capital Femoral Epiphyses; Coxa Vara; Femoral Neck Fractures

STUDY DESIGN:
Intervention Model Description: subtrochanteric valgus osteotomy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- subtrochanteric valgus osteotomy (Other): subtrochanteric valgus osteotomy
  Interventions: Procedure: subtrochanteric valgus osteotomy

INTERVENTIONS:
Procedure: subtrochanteric valgus osteotomy — subtrochanteric valgus osteotomy

SUMMARY:
Slipped Capital Femoral Epiphysis (SCFE) on Top of Fixed Fracture Neck of Femur managed by subtrochanteric valgus osteotomy

DETAILED DESCRIPTION:
The incidence of Slipped capital femoral epiphysis (SCFE) after management of femoral neck fracture in pediatrics is very rare. In this case report, a 9-year-old female child sustained left sided femur neck fracture after a motor car accident. The fracture was fixed by two cannulated screws and healing with mild varus occurred after 1.5 months. However, progressive slippage of femoral epiphysis was observed. This was treated by subtrochanteric valgus osteotomy

ELIGIBILITY:
Inclusion Criteria:

* scfe on top NOF

Exclusion Criteria:

* pathological fracture

Ages: 3 Years to 14 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
modified McKay's criteria | one year
  I excellent II Good III Fair IV Poor

SECONDARY OUTCOMES:
Rust union score | one year
  union
  1. absent callus visible fracture
  2. present callus visible fracture
  3. present callus invisible fracture

CONTACTS AND LOCATIONS:
Overall Officials: Hesaham M Elbaseet, MD, Principal Investigator — Assiut University
Locations (1):
- faculty of medicine Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yerli M, Ocak O, Yuce A, Bayraktar TO, Kir MC, Imren Y, Dedeoglu SS, Gurbuz H. Retrospective analysis of 35 pediatric femoral neck fractures. Eur J Orthop Surg Traumatol. 2022 Oct;32(7):1385-1390. doi: 10.1007/s00590-021-03126-6. Epub 2021 Sep 20. PMID 34542716
- [Background] Li H, Zhao L, Huang L, Kuo KN. Delayed Slipped Capital Femoral Epiphysis After Treatment of Femoral Neck Fracture in Children. Clin Orthop Relat Res. 2015 Aug;473(8):2712-7. doi: 10.1007/s11999-014-4067-y. Epub 2014 Nov 27. PMID 25427426